CLINICAL TRIAL: NCT01140685
Title: Analysis of Anti-inflammatory and Antioxidant Pathways in Lung Diseases by Haem Oxygenase-1 (HO-1) in Induced Sputum and Carbon Monoxide (CO) in Exhaled Air
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: ELIZABETH FIERMAN, PHD, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-10-LF-669-CTIL
Record Dates: First submitted 2010-02-17; First posted 2010-06-09 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-03

CONDITIONS: Lung Diseases
Keywords: mucus-stimulated (induced sputum); lung disease (asthma, COPD, ILD and OLD); HO-1 (heme oxigenase-1); oxidative stress; CO (carbon monoxide); The oxidative stress in lung diseases
MeSH Terms: conditions — Lung Diseases; Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — induced sputum, exhaled CO levels
Oversight: Data Monitoring Committee: No

SUMMARY:
This work will focus on the anti-inflammatory and antioxidant pathways in lung diseases by measuring HO-1 in induced sputum and CO in exhaled air in cases of four respiratory diseases, asthma, chronic obstructive pulmonary disease (COPD), occupational lung diseases (OLD) and interstitial lung disease (ILD).

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Ages >/= 18 years
* Diagnosed with one or more lung diseases
* Referred for sputum induction to the Pulmonary Laboratory in the Tel-Aviv Sourasky Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty adult male and female patients who had been diagnosed with one or more of the four study diseases and referred for sputum induction to the Pulmonary Laboratory in the Tel-Aviv Sourasky Medical Center will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
exhaled CO levels | 2010-2011

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Fierman, PHD, Principal Investigator — Tel Aviv Sorasky Medical Center